CLINICAL TRIAL: NCT00431847
Title: Regional Anesthesia in Combat Trauma Improves Pain Disability Outcomes
Brief Title: Regional Anesthesia Military Battlefield Pain Outcomes Study
Acronym: RAMBPOS
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); Brooke Army Medical Center (U.S. Federal Agency); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: D4506-I; NCT01710475 (obsolete NCT alias)
Record Dates: First submitted 2007-02-02; First posted 2007-02-06 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Anxiety Disorders; Complex Regional Pain Syndrome Type II; Depressive Disorders; Post-Traumatic Stress Disorder; Substance Abuse
Keywords: Anesthesia, Regional; Causalgia; Trauma; Complex Regional Pain Syndrome Type II; Neuropathic Pain; PTSD; Combat Stress Disorders; Afghan War, 2001-; Iraq War, 2003-
MeSH Terms: conditions — Anxiety Disorders; Causalgia; Depressive Disorder; Stress Disorders, Post-Traumatic; Substance-Related Disorders; Wounds and Injuries; Neuralgia; Combat Disorders | interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Soldiers with one or more severely injured, mangled or amputated limbs from the Iraq/Afghanistan war aggressively treated with regional anesthesia for pain control.
  Interventions: Procedure: Regional Anesthesia
- Group 2: Soldiers with one or more severely injured, mangled or amputated limbs from the Iraq/Afghanistan war receiving standard treatment for pain control.
  Interventions: Procedure: Standard Pain Management Protocol

INTERVENTIONS:
Procedure: Regional Anesthesia — Subject received regional anesthesia to affected limb(s) within 72 hours of traumatic event.
  Groups: Group 1
Procedure: Standard Pain Management Protocol — Intermittent dosing of analgesics and anxiolytics instituted prior to continuous intravenously dosing which was individually titrated to patient care goals.
  Other Names: No RA Group
  Groups: Group 2

SUMMARY:
The purpose of this study is to examine the short and long-term benefits of implementing early regional anesthesia techniques for pain control after a major traumatic injury to one or more extremities during combat in the Iraqi/Afghanistan war, including the effects on acute and chronic pain, quality of life, and mental health.

DETAILED DESCRIPTION:
BACKGROUND:

Adequate pain management for combat casualties balances the need for emergent, life-saving care with the urgency to remove soldiers from harm's way. Control of pain in traumatic battlefield situations may be impossible until safe evacuation to a surgical facility is achieved and a wounded soldier can receive general anesthesia. Recent evidence suggests that neural plasticity in the central nervous system coupled with hyperstimulation of central neuronal pathways lead to neuropathological remodeling. This neural rewiring may result in chronic pain for patients who have experienced severe, unrelieved acute pain. In addition, the stress of combat along with the suffering of prolonged uncontrolled pain may contribute to psychological disorders, such as post-traumatic stress disorder, depression, and substance abuse.

OBJECTIVE:

The purpose of this study is to evaluate the effect of early and aggressive advanced regional anesthesia on the chronic neuropathic pain, health related quality of life, and mental health of Operation Enduring Freedom (OEF) and Operation Iraqi Freedom (OIF) Veterans who have suffered a major limb injury in combat. An additional aim of this study is to quantify and characterize the short-term and long-term effects of traumatic combat limb injuries on post-injury acute pain, chronic pain, health related quality of life, functional status, social reintegration, psychological adjustment, and substance abuse behaviors in a population of injured military personnel.

METHOD:

This study employs a cohort repeated measures study design involving prospective data collection at scheduled intervals. Interviews with participants provide data on pain outcomes, psychiatric morbidities, and quality of life. Follow up evaluations conclude at the two year anniversary of the start of combat injury rehabilitation. Medical records information collected retrospectively from armed services treatment facilities provide data on the use of pain management therapies as well as individual responses to regional anesthesia.

IMPLICATIONS FOR RESULTS:

The findings of this study may impact the clinical field by providing information on the effectiveness and benefits of early advanced regional anesthesia for chronic pain control. This study may also provide data to determine whether regional anesthesia pain treatments prevent or reduce the development of psychological maladjustment disorders such as post-traumatic stress disorder, depression, and substance abuse in a population of military personnel with combat limb injuries.

ELIGIBILITY:
Inclusion Criteria:

* Major injury in one or more extremities requiring hospitalization and inpatient rehabilitation.

Exclusion Criteria:

* Major head trauma
* Cognitive deficits
* Inability to concentrate
* Poor judgment and impulse control
* Substantial hearing loss
* Bilateral upper extremity amputation with no alternate means to complete the survey forms

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Military service members with one or more severely injured, mangled or amputated limbs from Iraq/Afghanistan war.
Sampling Method: Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2007-10; Primary Completion 2013-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rollin M Gallagher, MD MPH, Principal Investigator — Pain Management Service
Locations (3):
- United States (3):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Pain Management Service, Philadelphia, Pennsylvania
  - Brooke Army Medical Center & US Army Institute of Surgical Research, Fort Sam Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gallagher RM, Polomano RC, Giordano NA, Farrar JT, Guo W, Taylor L, Oslin D, Goff BJ, Buckenmaier CC. Prospective cohort study examining the use of regional anesthesia for early pain management after combat-related extremity injury. Reg Anesth Pain Med. 2019 Sep 27:rapm-2019-100773. doi: 10.1136/rapm-2019-100773. Online ahead of print. PMID 31563880

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six hundred eighty-seven (687) combat-injured military service members hospitalized with at least one major limb injury were assessed for eligibility as an inpatient at one of two military treatment facilities. Three hundred one (301) of these patients did not meet criteria for study enrollment.
Pre-assignment Details: Three hundred eighty-six (386) participants provided study data. Twenty-Eight (28) of these participants were excluded from group observation due to completion of less than two study visits.
Groups:
- RA Within 7 Days From Injury: During initial hospital admission for combat injury, participant received standard pain management treatment which included first administration of regional anesthesia within seven days from the date of injury.
- RA 8 - 14 Days From Injury: During initial hospital admission for combat injury, participant received standard pain management treatment which included first administration of regional anesthesia at any point from day 8 to day 14 after date of injury.
- RA > 14 Days From Injury: During initial hospital admission for combat injury, participant received standard pain management treatment which included first administration of regional anesthesia greater than 14 days from the date of injury.
- No Regional Anesthesia (RA): During initial hospital admission for combat injury, participant received standard pain management treatment which did not include regional anesthesia.
- Unknown Treatment Status: No patient data on exposure to Regional Anesthesia
Period: Overall Study
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No Regional Anesthesia (RA) | Unknown Treatment Status
Started | 132 | 45 | 24 | 184 | 1
Completed | 126 (All participants with at least two study visits were included in analysis.) | 42 (All participants with at least two study visits were included in analysis.) | 20 (All participants with at least two study visits were included in analysis.) | 170 (All participants with at least two study visits were included in analysis.) | 0
Not Completed | 6 | 3 | 4 | 14 | 1
Not completed — completion of less than two study visits | 6 | 3 | 4 | 14 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No Regional Anesthesia (RA) | Total
Number analyzed (Participants) | 126 | 42 | 20 | 170 | 358
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.20 (6.30) | 26.68 (4.80) | 29.08 (8.97) | 28.15 (7.87) | 28.04 (7.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 2 | 3
  Male | 126 | 41 | 20 | 168 | 355
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 8 | 4 | 19 | 45
  Not Hispanic or Latino | 112 | 34 | 16 | 151 | 313
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 6 | 9
  Asian | 5 | 3 | 0 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 0 | 2 | 12 | 19
  White | 101 | 31 | 17 | 129 | 278
  More than one race | 12 | 6 | 1 | 17 | 36
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Education [Number; unit: participants]
  High School/GED | 47 | 18 | 8 | 74 | 147
  Some College | 47 | 18 | 9 | 72 | 146
  Bachelor's Degree or Higher | 32 | 6 | 3 | 24 | 65
Marital Status [Number; unit: participants]
  Never Married | 51 | 19 | 7 | 89 | 166
  Married or Living w/Partner | 70 | 22 | 13 | 67 | 172
  Separated/Divorced | 5 | 1 | 0 | 14 | 20
Number of Deployments, Continuous [Mean (Standard Deviation); unit: deployments] | 2.13 (1.27) | 1.80 (0.90) | 2.40 (2.54) | 1.85 (1.05) | 1.97 (1.25)
Injury Severity Score (ISS) [Mean (Standard Deviation); unit: units on a scale] — Injury Severity Scores (ISS): ISS is a scale to evaluate anatomic injury severity following trauma that ranges from 0 to 75, with 75 indicating the greatest severity. An Abbreviated Injury Scale (AIS) score is allocated to the six body regions (Head, Face, Chest, Abdomen, Extremities, and External). The highest AIS score in each body region is used. The 3 most severely injured body regions scores are squared and summed to produce the ISS. The ISS correlates linearly with mortality, morbidity, and hospital stay.
  units on a scale | 17.31 (8.56) | 19.74 (11.88) | 24.65 (12.59) | 18.07 (11.57) | 18.37 (10.79)
Length of Initial Hospital Stay [Mean (Standard Deviation); unit: months] | 41.14 (30.54) | 47.45 (33.74) | 59.90 (47.64) | 27.95 (30.72) | 36.69 (33.35)

OUTCOME MEASURES:

1. Primary Outcome: Neuropathic Pain Scale - Pain Intensity
Description: The Neuropathic Pain Scale (NPS) is a 10-item self-report questionnaire designed to assess the distinct pain qualities associated with neuropathic pain, pain initiated or caused by a dysfunction of the nervous system. Item numbers ask respondents to describe the intensity of their combat limb pain on a scale of 0 - 10, where "0" is no pain and "10" is the most intense pain imaginable.
Time Frame: Means of the individuals aggregated to the cohort level from start of rehabilitation for combat injury, month 0, to end of study follow up, at 30 months
Measure: Mean (Standard Error); unit: units on the Neuropathic Pain Scale
Groups:
- No RA: During initial hospital admission for combat injury, participant received standard pain management treatment which did not include regional anesthesia.
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on the Neuropathic Pain Scale | 3 (0.16) | 3.44 (0.3) | 3.92 (0.45) | 3.04 (0.15)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; A Linear Mixed Effects Model is utilized to examine the longitudinal progression of each outcome related to RA administration while adjusting for injury severity and length of stay of initial hospitalization for injury. The main treatment effect (RA group) is treated as a classification variable with the No RA group used as the reference group. The overall slope of the model (below) is reported as a continuous variable for time since injury; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Slope = -0.03230, 95% CI 2-sided [-0.0448 to -0.02013], Standard Error of Mean 0.006190
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; A Linear Mixed Effects Model is utilized to examine the longitudinal progression of each outcome related to RA administration while adjusting for injury severity and length of stay of initial hospitalization for injury. The time interaction component of the model is reported below; Test type: Superiority or Other; p = 0.4492, Chi-squared; Degrees of Freedom: 3; Chi Squared = 2.65
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; A Linear Mixed Effects Model is utilized to examine the longitudinal progression of each outcome related to RA administration while adjusting for injury severity and length of stay of initial hospitalization for injury. The main treatment effect (RA group) is treated as a classification variable with the No RA group used as the reference group; Test type: Superiority or Other; p = 0.640, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -0.1080, 95% CI 2-sided [-0.5621 to 0.3461], Standard Error of Mean 0.2308 — Estimated intercept group difference
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.3286, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.3299, 95% CI 2-sided [-0.3334 to 0.9932], Standard Error of Mean 0.3372
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0694, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.8591, 95% CI 2-sided [-0.06841 to 1.7866], Standard Error of Mean 0.4716

2. Primary Outcome: Neuropathic Pain Scale - Overall Pain Quality
Description: The Neuropathic Pain Scale (NPS) is a 10-item self-report questionnaire designed to assess the distinct pain qualities associated with neuropathic pain, pain initiated or caused by a dysfunction of the nervous system. The NPS Overall Pain Quality composite score is a measure of six distinct pain qualities of respondents' combat limb pain on a scale of 0 - 10, where "0" is no pain and "10" is the most intense sensation imaginable. The six pain qualities included in the composite score is sharp, hot, dull, cold, itchy, and sensitive to touch.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on the Neuropathic Pain Scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on the Neuropathic Pain Scale | 1.90 (0.11) | 2.04 (0.20) | 2.13 (0.27) | 1.82 (0.10)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Slope = -0.02332, 95% CI 2-sided [-0.03076 to -0.01589], Standard Error of Mean 0.003777
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.4772, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 2.49
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.6077, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.07724, 95% CI 2-sided [-0.2184 to 0.3729], Standard Error of Mean 0.1503
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.3616, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.2004, 95% CI 2-sided [-0.2311 to 0.6319], Standard Error of Mean 0.2194
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.3155, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.3082, 95% CI 2-sided [-0.2948 to 0.9112], Standard Error of Mean 0.3066

3. Primary Outcome: Neuropathic Pain Scale - Total Score
Description: The Neuropathic Pain Scale (NPS) is a 10-item self-report questionnaire designed to assess the distinct pain qualities associated with neuropathic pain, pain initiated or caused by a dysfunction of the nervous system. It has a scale of 0 - 10, where "0" is no pain and "10" is the most intense sensation imaginable. The NPS total score is an average of all ten items.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on the Neuropathic Pain Scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on the Neuropathic Pain Scale | 2.35 (0.12) | 2.60 (0.22) | 2.80 (0.31) | 2.29 (0.11)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Slope = -0.02746, 95% CI 2-sided [-0.03573 to -0.01919], Standard Error of Mean 0.004202
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3345, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 3.40
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.8223, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.03860, 95% CI 2-sided [-0.2993 to 0.3765], Standard Error of Mean 0.1718
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.2448, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.2919, 95% CI 2-sided [-0.2009 to 0.7848], Standard Error of Mean 0.2506
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.2014, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.4482, 95% CI 2-sided [-0.2405 to 1.1369], Standard Error of Mean 0.3502

4. Primary Outcome: Brief Pain Inventory - Worst Pain
Description: The Brief Pain Inventory - Short form (BPI) is a 17-item self-report questionnaire designed to assess severity of pain and the degree to which pain interferes with common dimensions of feeling and function. BPI Item - Worst Pain asks the respondent to rate worst pain in the past week from the combat limb injury on a scale of 0 to 10, where "0" is no pain, and "10" is pain as bad as you can imagine.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on the Brief Pain Inventory Scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on the Brief Pain Inventory Scale | 4.54 (0.18) | 4.95 (0.36) | 5.83 (0.44) | 4.62 (0.19)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Slope = -0.04030, 95% CI 2-sided [-0.5446 to -0.02613], Standard Error of Mean 0.007196
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3631, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 3.19
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.7148, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -0.1004, 95% CI 2-sided [-0.6404 to 0.4396], Standard Error of Mean 0.2746
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.3741, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.3568, 95% CI 2-sided [-0.4318 to 1.1453], Standard Error of Mean 0.4009
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0213, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 1.2969, 95% CI 2-sided [0.1938 to 2.4000], Standard Error of Mean 0.5609

5. Primary Outcome: Brief Pain Inventory - Average Pain
Description: The Brief Pain Inventory - Short form (BPI) is a 17-item self-report questionnaire designed to assess severity of pain and the degree to which pain interferes with common dimensions of feeling and function. BPI Item - Average Pain asks the respondent to rate combat limb injury pain on average (no time frame given) on a scale of 0 to 10, where "0" is no pain, and "10" is pain as bad as you can imagine.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on the Brief Pain Inventory Scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on the Brief Pain Inventory Scale | 2.18 (0.13) | 2.45 (0.23) | 3.21 (0.42) | 2.45 (0.13)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Slope = -0.02776, 95% CI 2-sided [-0.03702 to -0.01850], Standard Error of Mean 0.004706
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2752, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 3.88
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.1094, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -0.3079, 95% CI 2-sided [-0.6851 to 0.06941], Standard Error of Mean 0.1918
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.8786, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.0428, 95% CI 2-sided [-0.5079 to 0.5935], Standard Error of Mean 0.2800
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0847, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.6759, 95% CI 2-sided [-0.09297 to 1.4448], Standard Error of Mean 0.3910

6. Primary Outcome: Brief Pain Inventory - Pain Interference
Description: The Brief Pain Inventory - Short form (BPI) is a 17-item self-report questionnaire designed to assess severity of pain and the degree to which pain interferes with common dimensions of feeling and function. The BPI measures how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. BPI pain interference is scored as the mean of the seven interference items, each ranging 0 to 10, where "0" is pain from combat limb injury does not interfere and "10" is pain from combat limb injury completely interferes with this aspect of daily life.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on the Brief Pain Inventory Scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on the Brief Pain Inventory Scale | 1.91 (0.15) | 2.03 (0.25) | 2.57 (0.46) | 1.88 (0.14)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Slope = -0.03645, 95% CI 2-sided [-0.04808 to -0.02481], Standard Error of Mean 0.005913
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3677, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 3.16
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.7926, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -0.05816, 95% CI 2-sided [-0.4929 to 0.3766], Standard Error of Mean 0.2210
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.5953, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.1708, 95% CI 2-sided [-0.4610 to 0.8026], Standard Error of Mean 0.3212
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.1261, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.6873, 95% CI 2-sided [-0.1943 to 1.5689], Standard Error of Mean 0.4482

7. Primary Outcome: Brief Pain Inventory - Treatment Relief
Description: The Brief Pain Inventory - Short form (BPI) is a 17-item self-report questionnaire designed to assess the severity of pain and the degree to which pain interferes with common dimensions of feeling and function. The BPI measures in the last 24 hours, how much relief pain treatments or medications provided on a scale of 0%, meaning no relief, to 100%, indicating complete relief.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of pain relief
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
percentage of pain relief | 67.53 (2.39) | 66.80 (3.04) | 58.58 (4.88) | 66.77 (1.86)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Slope = -0.4831, 95% CI 2-sided [-0.7286 to -0.2377], Standard Error of Mean 0.1243
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3617, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 3.20
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.2532, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 3.1574, 95% CI 2-sided [-2.2715 to 8.5863], Standard Error of Mean 2.7573
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.7580, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 1.2227, 95% CI 2-sided [-6.5833 to 9.0286], Standard Error of Mean 3.9633
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.1837, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -7.1649, 95% CI 2-sided [-17.7484 to 3.4187], Standard Error of Mean 5.3759

8. Primary Outcome: SF-36 Physical Component Summary
Description: The Physical component score (PCS) is an aggregate of the eight subscale scores measuring physical components with each subscale ranging from worst possible health, 0, to 100, the highest possible score and therefore the optimal health state. After the eight scale scores are calculated, a z-score is calculated for each by subtracting the scale mean of a sample of the U.S. general population from an individual's scale score and then dividing by the standard deviation from the U.S. general population. Each of the eight z-scores is then multiplied by the corresponding factor scoring coefficient for the scale. The products of the z-scores and factor scoring coefficients for the PCS are then summed together. Each resulting sum is multiplied by 10 and added to 50 to linearly transform the PCS to the T-score metric, which has a mean of 50 and a standard deviation of 10 for the U.S. general population (Taft et al., 2001) doi:10.1023/A:1012552211996
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: t-score
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
t-score | 40.30 (0.96) | 37.00 (1.72) | 31.51 (2.05) | 41.94 (0.92)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Slope = 0.4741, 95% CI 2-sided [0.3971 to 0.5511], Standard Error of Mean 0.03909
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6075, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 1.83
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.4558, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -0.9534, 95% CI 2-sided [-3.4675 to 1.5607], Standard Error of Mean 1.2763
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0914, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -3.3505, 95% CI 2-sided [-7.2442 to 0.5432], Standard Error of Mean 1.9770
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -8.3700, 95% CI 2-sided [-14.4589 to -2.2810], Standard Error of Mean 3.0921

9. Primary Outcome: SF-36 Mental Component Summary
Description: The Mental component score (MCS) is an aggregate of the eight subscale scores that account for measuring physical components with each subscale ranging from worst possible health, 0, to 100, the highest possible score and therefore the optimal health state. After the eight scale scores are calculated, a z-score is determined for each by subtracting the scale mean of a sample of the U.S. general population from an individual's scale score and then dividing by the standard deviation from the U.S. general population. Each of the eight z-scores is then multiplied by the corresponding factor scoring coefficient for the scale. The products of the z-scores and factor scoring coefficients for the MCS are then summed together. Each resulting sum is multiplied by 10 and added to 50 to linearly transform the MCS to the T-score metric, which has a mean of 50 and a standard deviation of 10 for the U.S. general population (Taft et al., 2001) doi:10.1023/A:1012552211996
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: t-score
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
t-score | 52.47 (1.11) | 52.12 (1.84) | 49.90 (2.94) | 51.30 (0.82)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Slope = -0.2169, 95% CI 2-sided [-0.2987 to -0.1352], Standard Error of Mean 0.04148
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0950, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 6.37
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.5878, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.7246, 95% CI 2-sided [-1.9056 to 3.3547], Standard Error of Mean 1.3351
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.9053, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -0.2466, 95% CI 2-sided [-4.3231 to 3.8299], Standard Error of Mean 2.0697
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.4682, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -2.3457, 95% CI 2-sided [-8.7034 to 4.0120], Standard Error of Mean 3.2285

10. Primary Outcome: Post Traumatic Stress Disorder (PTSD) Total Severity
Description: Post-Traumatic Stress Disorder Checklist (PCL): The PCL is a 17-item PTSD assessment instrument that asks respondents to rate the extent to which they have experienced each of the 17 diagnostic symptoms for PTSD outlined in the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV). Scores are computed by adding the 17 items scored 1 to 5. Scores range from 17 to 85. Higher scores indicate higher severity of symptoms.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on the PCL scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on the PCL scale | 27.99 (1.10) | 30.23 (1.98) | 25.62 (2.00) | 27.63 (0.87)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1938, Mixed Models Analysis; Slope = 0.04639, 95% CI 2-sided [-0.02369 to 0.1165], Standard Error of Mean 0.03562
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.4884, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 2.43
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.6593, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 0.6174, 95% CI 2-sided [-2.1348 to 3.3696], Standard Error of Mean 1.3991
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0889, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 3.4575, 95% CI 2-sided [-0.5280 to 7.4431], Standard Error of Mean 2.0263
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.8727, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -0.4499, 95% CI 2-sided [-5.9692 to 5.0694], Standard Error of Mean 2.8061

11. Primary Outcome: Treatment Outcomes in Pain Survey (TOPS): Fear Avoidance
Description: Treatment Outcomes in Pain Survey (TOPS): The 112-item TOPS explicitly acknowledges and measures contextual factors that are important in pain treatment including the dimensions of pain symptoms, fear avoidance, patient satisfaction with outcomes, and health care satisfaction. TOPS scoring ranges from 100, the worst possible score where pain impacts all components of the health domain, to 0, the best possible response where pain does not interfere with any component in the domain.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on TOPS scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on TOPS scale | 41.85 (2.07) | 43.57 (3.65) | 51.27 (6.29) | 40.62 (1.91)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; Slope = -0.5230, 95% CI 2-sided [-0.6973 to -0.3486], Standard Error of Mean 0.08855
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1800, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 4.89
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.4151, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 2.3020, 95% CI 2-sided [-3.2530 to 7.8570], Standard Error of Mean 2.8198
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.3157, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 4.3376, 95% CI 2-sided [-4.1592 to 12.8344], Standard Error of Mean 4.3140
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0911, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 11.8250, 95% CI 2-sided [-1.9040 to 25.5541], Standard Error of Mean 6.9715

12. Primary Outcome: Treatment Outcomes in Pain Survey (TOPS): Health Care Satisfaction
Description: Treatment Outcomes in Pain Survey (TOPS): The 112-item TOPS explicitly acknowledges and measures contextual factors that are important in pain treatment including the dimensions of pain symptoms, fear avoidance, patient satisfaction with outcomes, and health care satisfaction. For the health care satisfaction scale of the TOPS, scoring ranges from 100, the best possible score where satisfaction is optimal, to 0, least satisfied.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on TOPS scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on TOPS scale | 61.01 (1.80) | 56.29 (3.54) | 47.68 (4.67) | 58.77 (1.68)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; Slope = -0.2888, 95% CI 2-sided [-0.4675 to -0.1100], Standard Error of Mean 0.09078
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0966, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 6.33
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.2195, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 2.9879, 95% CI 2-sided [-1.7938 to 7.7697], Standard Error of Mean 2.4264
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.5105, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -2.4636, 95% CI 2-sided [-9.8289 to 4.9018], Standard Error of Mean 3.7381
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0903, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -10.3871, 95% CI 2-sided [-22.4174 to 1.6433], Standard Error of Mean 6.1087

13. Primary Outcome: Treatment Outcomes in Pain Survey (TOPS):Life Control
Description: as for outcome 11
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on TOPS scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on TOPS scale | 75.82 (1.92) | 68.02 (4.15) | 58.52 (5.76) | 73.76 (1.70)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6602, Mixed Models Analysis; Slope = -0.04113, 95% CI 2-sided [-0.2252 to 0.1429], Standard Error of Mean -0.04113
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6764, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 1.53
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.3458, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 2.4902, 95% CI 2-sided [-2.7036 to 7.6840], Standard Error of Mean 2.6357
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.1969, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -5.2518, 95% CI 2-sided [-13.2466 to 2.7430], Standard Error of Mean 4.0583
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0480, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -12.9796, 95% CI 2-sided [-25.8429 to -0.1162], Standard Error of Mean 6.5287

14. Primary Outcome: Treatment Outcomes in Pain Survey (TOPS): Observed Family Social Disability
Description: as for outcome 11
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on TOPS scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on TOPS scale | 48.29 (2.37) | 51.04 (4.05) | 57.51 (4.33) | 47.87 (1.75)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0199, Mixed Models Analysis; Slope = -0.2349, 95% CI 2-sided [-0.4323 to -0.03745], Standard Error of Mean 0.1003
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.4577, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 2.60
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.7417, Mixed Models Analysis; Mean Difference (Net) = -0.9502, 95% CI 2-sided [-6.6240 to 4.7236], Standard Error of Mean 2.8797
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.7778, Mixed Models Analysis; Mean Difference (Net) = 1.2580, 95% CI 2-sided [-7.5129 to 10.0289], Standard Error of Mean 4.4523
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.2411, Mixed Models Analysis; Mean Difference (Net) = 8.5232, 95% CI 2-sided [-5.7608 to 22.8073], Standard Error of Mean 7.2532

15. Primary Outcome: Treatment Outcomes in Pain Survey (TOPS): Patient Satisfaction With Outcomes
Description: Treatment Outcomes in Pain Survey (TOPS): The 112-item TOPS explicitly acknowledges and measures contextual factors that are important in pain treatment including the dimensions of pain symptoms, fear avoidance, patient satisfaction with outcomes, and health care satisfaction. For the satisfaction with outcomes scale of the TOPS, scoring ranges from 100, the best possible score where satisfaction is optimal, to 0, least satisfied.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on TOPS scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on TOPS scale | 66.72 (1.75) | 61.46 (3.56) | 53.06 (5.00) | 66.24 (1.67)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0504, Mixed Models Analysis; Slope = 0.1629, 95% CI 2-sided [-0.00029 to 0.3261], Standard Error of Mean 0.08284
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6942, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 1.45
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.5297, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 1.5241, 95% CI 2-sided [-3.2469 to 6.2951], Standard Error of Mean 2.4216
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.3155, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -3.7679, 95% CI 2-sided [-11.1478 to 3.6120], Standard Error of Mean 3.7464
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.1105, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -9.7558, 95% CI 2-sided [-21.7515 to 2.2399], Standard Error of Mean 6.0920

16. Primary Outcome: Treatment Outcomes in Pain Survey (TOPS): Pain Symptoms
Description: as for outcome 11
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on TOPS scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on TOPS scale | 35.97 (1.92) | 41.22 (3.86) | 48.82 (5.91) | 36.80 (1.77)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Slope = -.2979, 95% CI 2-sided [-0.4465 to -0.1493], Standard Error of Mean 0.07538
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.4361, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 2.72
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.7297, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -0.9001, 95% CI 2-sided [-6.0247 to 4.2246], Standard Error of Mean 2.6015
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.2868, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 4.2896, 95% CI 2-sided [-3.6250 to 12.2043], Standard Error of Mean 4.0186
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.1516, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 9.0118, 95% CI 2-sided [-3.3270 to 21.3505], Standard Error of Mean 6.2663

17. Primary Outcome: Treatment Outcomes in Pain Survey (TOPS): Solicitous Responses
Description: as for outcome 11
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on TOPS scale
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No RA
Number analyzed (Participants) | 126 | 42 | 20 | 170
units on TOPS scale | 48.29 (2.37) | 51.07 (5.18) | 71.65 (6.85) | 48.02 (2.57)
Statistical Analysis 1: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; A Linear Mixed Effects Model is utilized to examine the longitudinal progression of each outcome related to RA administration while adjusting for injury severity and length of stay of initial hospitalization for injury. The main treatment effect (RA group) is treated as a classification variable with the No RA group used as the reference group. The overall slope of the model (below) is reported as a continuous variable for time since injury. T; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Slope = -0.9776, 95% CI 2-sided [-1.2584 to -0.6967], Standard Error of Mean 0.1426
Statistical Analysis 2: Comparison: RA Within 7 Days From Injury vs RA 8 - 14 Days From Injury vs RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8548, Chi-squared; Degrees of Freedom: 3; Chi-Squared = 0.78
Statistical Analysis 3: Comparison: RA Within 7 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.3882, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 3.3635, 95% CI 2-sided [-4.3026 to 11.0296], Standard Error of Mean 3.8899
Statistical Analysis 4: Comparison: RA 8 - 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.9322, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = -0.5029, 95% CI 2-sided [-12.1376 to 11.1317], Standard Error of Mean 5.9044
Statistical Analysis 5: Comparison: RA > 14 Days From Injury vs No RA; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0233, Mixed Models Analysis; RA groups treated as classification variables with No RA group as reference; Mean Difference (Net) = 21.1166, 95% CI 2-sided [2.8992 to 39.3341], Standard Error of Mean 9.2462

ADVERSE EVENTS:
Time Frame: 0, 1, 2, 3, 4, 5, 6, 9, 12, 15, 18, and 24 months after start of injury rehabilitation
Arm/Group | RA Within 7 Days From Injury | RA 8 - 14 Days From Injury | RA > 14 Days From Injury | No Regional Anesthesia (RA)
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/42 | 0/20 | 0/170
Other Adverse Events (participants affected / at risk) | 0/126 | 0/42 | 0/20 | 0/170

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No